CLINICAL TRIAL: NCT06687629
Title: Best Practice in the Management of Concha Bullosa in FESS Operation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Mario Järvekülg, specialist doctor, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUS/66/2018
Record Dates: First submitted 2024-11-12; First posted 2024-11-13 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-10

CONDITIONS: Sinusitis; Sinusitis Bacterial; Sinusitis Recurrent; Turbinate; Hypertrophy Mucous Membrane; Turbinate Hypertrophy; Concha Bullosa; Middle Turbinate
Keywords: concha bullosa; sinusitis; concha bullosa resection; concha bullosa crushing; chronic sinusitis; sinusitis bacterial
MeSH Terms: conditions — Sinusitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- crushing (Active Comparator): Concha bullosa crushing group
  Interventions: Procedure: Concha bullosa crushing
- resection (Active Comparator): Concha bullosa resection group
  Interventions: Procedure: Concha bullosa resection

INTERVENTIONS:
Procedure: Concha bullosa crushing — Concha bullosa crushing
  Arms: crushing
Procedure: Concha bullosa resection — Concha bullosa resection
  Arms: resection

SUMMARY:
Concha bullosa (CB) refers to the condition where the middle turbinate's interior is aerated (making the turbinate wide and thick). CB can narrow the middle meatus and the ostiomeatal complex. In adults suffering from chronic sinusitis, the prevalence of CB is approximately 34%. The most common treatment method for CB is turbinate crushing. This is considered a conservative treatment that preserves the mucous membranes relatively intact without opening the interior of the turbinate. Another fairly common method is the removal of the lateral part of the bullous middle turbinate. Opening the CB and removing the lateral part of the middle turbinate can lead to adhesions between the middle turbinate and the lateral wall of the nose. These adhesions can impede airflow and narrow or completely close the ostium or the surgically created middle meatal antrostomy. Crushing the CB is technically easier and possibly a less traumatic procedure. However, it is suspected that some of these crushed bullous turbinates may refill. The development of a mucocele is another potential issue. Crushing might be a better option compared to resection in the long term. Preserving the mucous membranes during crushing may reduce the formation of adhesions, which are sometimes seen after resection of the middle turbinate. The purpose of the study is to investigate the long-term benefits and side effects of CB treatment methods. The study will include 60 patients undergoing a basic Functional Endoscopic Sinus Surgery (FESS) procedure due to recurrent or chronic maxillary sinusitis. The patients will be randomized, with 31 undergoing resection and 31 undergoing crushing. Before the procedure, patients will undergo a CT scan (NSO-TT) and symptom evaluation through various questionnaires. All patients will also undergo nasoscopy.

One year after the procedure, the patients' conditions will be reassessed (questionnaires, nasoscopy, NSO-TT only if necessary), including the need for revision surgery.

ELIGIBILITY:
Inclusion Criteria:

* chronic or recurrent rhinosinusitis
* 3 months of regular nasal corticosteroid usage
* No prior endoscopic procedures of the paranasal sinuses
* EPOS criteria for CRS are met: inflammation of the paranasal sinuses with at least 2 symptoms, one of which must be nasal obstruction/congestion or nasal discharge (anterior/posterior):

  * facial pain/pressure in the facial area
  * reduced or lost sense of smell SNOT-22 25 or higher

    * Complications of CRS (e.g., mucocele)
    * Pregnancy/breastfeeding or plans for them in the near future
    * Coagulation disorders
    * Systemic diseases: cystic fibrosis, primary ciliary dysfunction, sarcoidosis, Wegener's granulomatosis
    * Immunosuppression: diagnosed SAD, CVI, HIV, or use of biological/immunosuppressive drugs
    * Immunotherapy
    * Daily use of systemic corticosteroids
    * Communication issues (non-Finnish-speaking patient, neurological/psychiatric problems)
    * SNOT-22 score < 25

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2018-03-21 (Actual); Primary Completion 2023-07-12 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
postoperative SNOT-22 | 1 year
  postoperative SNOT-22 score

SECONDARY OUTCOMES:
LM endoscopy score | 1 year
  LM endoscopy score

OTHER OUTCOMES:
Antibiotics usage postoperatively | 1 year
  Antibiotics usage postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Markus Lilja, PhD, Study Director — Helsinki University Central Hospital; Mario Järvekülg, MD, Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Helsinki University Hospital Ear Clinic, Helsinki, Uusimaa, Finland

IPD SHARING:
Plan to Share IPD: No
According to the data protection regulations, patients' personal data cannot be shared publicly in Finland.

REFERENCES:
- [Background] Dogru H, Uygur K, Tuz M. Concha bullosa squeezer for turbinoplasty (Dogru forceps). J Otolaryngol. 2004 Apr;33(2):111-3. doi: 10.2310/7070.2004.02112. No abstract available. PMID 15518100